CLINICAL TRIAL: NCT07343323
Title: A Randomized, Single Center, Double-blind, Placebo-controlled, First in Human Study With Single Ascending Doses to Determine Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous Infusion and Subcutaneous Injections of KINE-101 in Healthy Subjects
Brief Title: A First-in-Human Study of KINE-101 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kine Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA101-CR3-001
Record Dates: First submitted 2025-12-10; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KINE-101 (Experimental)
  Interventions: Drug: KINE-101
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KINE-101 — KINE-101 injection, 12.5 mg/mL, administered once either intravenously (10 mg, 30 mg, 100 mg, or 300 mg) or subcutaneously (96.8 mg) on Day 1, depending on cohort.
  Arms: KINE-101
Drug: Placebo — Sterile 0.9% sodium chloride solution, administered once intravenously or subcutaneously on Day 1, matching the route of the investigational product.
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single ascending dose (SAD) study that evaluates the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of intravenous (IV) and subcutaneous (SC) formulations of KINE-101 in healthy volunteers at a single study center. Five cohorts of eight subjects each (six receiving KINE-101 and two receiving placebo) are admitted on Day -1, receive a single dose of investigational medicinal product (IMP) on Day 1, and remain in-house until Day 3, followed by outpatient visits on Days 7, 14, 28, and 42. Sentinel dosing applies in the first sub-cohort of each cohort: two sentinel subjects are dosed at least 10 minutes apart, and if no safety concerns arise during the 48-hour post-dose evaluation period, the remaining subjects in the cohort are subsequently dosed. Dosing in the second sub-cohort also occurs at intervals of at least 10 minutes. Four cohorts receive the IV formulation, with doses escalating from 10 mg up to an anticipated maximum of 300 mg. To compare relative bioavailability and characterize PK after subcutaneous administration, one SC cohort receives a single 96.8 mg dose. The number of cohorts and dose progression depend on emerging safety and PK data. Decisions to escalate, repeat, or modify dose levels are made by the Safety Review Committee (SRC), and additional cohorts may be added if deemed necessary.

ELIGIBILITY:
Inclusion Criteria:

* Signed IRB-approved informed consent before any screening procedures.
* Healthy subjects with no clinically significant illness or disease based on medical history, physical exam, ECG, and lab tests.
* Males and females aged 18-55 years at screening.
* Nonsmokers or no nicotine use for ≥1 year; urine cotinine <200 ng/mL at screening and admission.
* BMI 18.5-30.0 kg/m² and body weight ≥50 kg at screening.
* Suitable veins for venipuncture/cannulation.
* Able to fast overnight (≥10 hours).
* Male subjects agree to use condoms during intercourse and for 1 month after last IMP dose.
* Male subjects must not donate sperm from dosing day until 1 month after last IMP dose.
* Female subjects must be of non-childbearing potential (postmenopausal ≥12 months with FSH >40 IU/L or surgical sterilization such as hysterectomy, tubal ligation, bilateral oophorectomy/salpingectomy).

Exclusion Criteria:

* Received an investigational medicinal product (IMP) within 30 days or 5× half-life before first IMP administration.
* History of alcohol abuse within 2 years, weekly intake >21 units, or positive alcohol test at screening/admission.
* Current smokers or nicotine use within 12 months; positive urine cotinine at screening/admission.
* Clinically significant abnormal labs: ALT, AST, or total bilirubin >ULN (or >1.5×ULN if Gilbert's), serum creatinine >ULN, eGFR <80 mL/min/1.73 m², abnormal TSH, or other clinically relevant abnormal values.
* Positive drug abuse test at screening or admission.
* Positive HBsAg, anti-HCV, or HIV antibody at screening.
* Clinically significant psychiatric, cardiovascular, renal, hepatic, or chronic respiratory disease, including arrhythmia.
* Supine BP <90 or >140 mmHg systolic, or <50 or >90 mmHg diastolic after 5 minutes supine.
* Supine pulse <50 bpm or >100 bpm after 5 minutes supine.
* Personal or family history of long QTc syndrome, sudden cardiac death, or hERG mutation.
* Severe adverse reaction or hypersensitivity to any drug or excipients.
* Blood donation or loss >400 mL within 3 months or hemoglobin below normal limits.
* Use of prohibited medications, OTC drugs, herbal remedies, or supplements within 28 days before IMP administration.
* Received live or attenuated vaccines or systemic corticosteroids within 3 months prior to first IMP dose.
* Conditions interfering with drug absorption, distribution, metabolism, or excretion.
* Employees of sponsor/CRO or close relatives involved in the study.
* Unable to communicate meaningfully with study staff.
* QTcF >450 ms at screening or admission.
* Significant liver impairment or abnormal conjugated/direct bilirubin >ULN.
* Consumption of methylxanthines (tea, coffee, chocolate), quinine-containing drinks, grapefruit, Seville oranges, poppy seeds, or alcohol within protocol-defined windows before IMP administration.
* Investigator judges subject unfit for any reason.
* Positive SARS-CoV-2 RT-PCR within 4 weeks prior to screening.
* COVID-19 symptoms within 14 days prior to screening.
* Severe COVID-19 history (e.g., ECMO, mechanical ventilation).
* Unable to attend in-person visits per site COVID guidelines.
* Scheduled to receive COVID-19 vaccination within 2 weeks before or after IMP administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Day 1 to Day 42
  Incidence, severity, and relationship of treatment-emergent adverse events following single ascending doses of KINE-101.
Number of Participants with Clinically Significant Abnormal Hematology | Day 1 to Day 42
  Count of participants with clinically significant abnormal hematology findings (e.g., white blood cell count, hemoglobin, platelet count), as defined per protocol.
Number of Participants with Clinically Significant Abnormal Clinical Chemistry | Day 1 to Day 42
  Count of participants with clinically significant abnormal clinical chemistry findings (e.g., ALT, AST, creatinine), as defined per protocol.
Number of Participants with Clinically Significant Abnormal Urinalysis | Day 1 to Day 42
  Count of participants with clinically significant abnormal urinalysis findings (e.g., bilirubin, glucose, pH and specific gravity), as defined per protocol.
Number of Participants with Clinically Significant Abnormal Vital Signs | Day 1 to Day 42
  Count of participants with clinically significant abnormal vital sign findings (e.g., systolic and diastolic blood pressure, pulse, body temperature, respiratory rate), as defined per protocol.
Number of Participants with Clinically Significant Abnormal Electrocardiogram | Day 1 to Day 42
  Count of participants with clinically significant abnormal 12-lead electrocardiogram findings (e.g., PR interval, QRS interval, QT interval), as defined per protocol.
Number of Participants with Clinically Significant Abnormal Physical Examination | Day 1 to Day 42
  Count of participants with clinically significant abnormal physical examination findings, as defined per protocol.
Local Tolerability and Injection/Infusion Site Reactions | Day 1 to Day 42
  Local tolerability and pain assessed using the Numerical Rating Scale (NRS; 0 = no pain, 10 = worst possible pain). Higher scores indicate worse outcomes, as defined per protocol.

SECONDARY OUTCOMES:
Peak Plasma Concentration of KINE-101 (Cmax) | From predose on Day 1 through 24 hours postdose (Day 2)
  Maximum observed plasma concentration of KINE-101.
Time to Peak Plasma Concentration of KINE-101 (Tmax) | From predose on Day 1 through 24 hours postdose (Day 2)
  Time to reach the maximum observed plasma concentration of KINE-101.
Area Under the Plasma Concentration-Time Curve to Last Quantifiable Concentration (AUClast) | From predose on Day 1 through 24 hours postdose (Day 2)
  Area under the plasma concentration-time curve of KINE-101 from predose to the time of the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve Over the Dosing Interval (AUCtau) | From predose on Day 1 through 24 hours postdose (Day 2)
  Area under the plasma concentration-time curve of KINE-101 from predose over the dosing interval following single ascending doses.
Area Under the Plasma Concentration-Time Curve Extrapolated to Infinity (AUCinf) | From predose on Day 1 through 24 hours postdose (Day 2)
  Area under the plasma concentration-time curve of KINE-101 from predose extrapolated to infinite time.

OTHER OUTCOMES:
Pharmacodynamics of KINE-101 following single ascending doses | From predose on Day 1 through Day 28
  Pharmacodynamic assessments include changes from baseline in cytokines (such as IL-6, IL-10, CXCL13, IgM, IgG) and immunophenotyping markers (such as CD4+, CD25+, FoxP3+, CD39high, CTLA-4+, CD69+) to evaluate target engagement and explore PK/PD relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Park, Study Director — Kine Sciences Co., Ltd.
Locations (1):
- Parexel International, Baltimore, Maryland, United States